CLINICAL TRIAL: NCT00852150
Title: Reproducibility of Modified Lanza Scale for the Reporting of Gastritis and Duodenitis
Brief Title: Is a Reporting System for Gastritis or Duodenitis (Modified Lanza Scale) Reproducible?
Status: Completed | Type: Observational
Sponsor: Ruttonjee Hospital (Other)
Responsible Party: Principal Investigator, Fook-Hong Ng, SMO, Ruttonjee Hospital
Other Study IDs: HKEC 2008-083
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Gastritis; Duodenitis
Keywords: gastritis; duodenitis; inter-rater reliability; intra-rater reliablity; gastroscopy; duodenoscopy
MeSH Terms: conditions — Gastritis; Duodenitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The modified Lanza scale (Lanza FL, 1984) has been widely utilized to grade the degree of gastritis and duodenitis. However, the inter-rater or intra-rater reproducibility of this scale has never been validated. As a quality improvement program, it is important to study the reproducibility of the scale between different operators and the operators himself.

Method: During upper endoscopic examinations, one investigator performed the procedure and the second investigator look at the endoscopic image. The degree of gastritis and duodenitis is graded. The results of the grading are blinded to the other investigator.

The endoscopic video is stored for reassessment to determine the intra-rater reliability. The patient identifier is stored in serial number. The investigator will not retrieve the report of the first assessment during the second assessment.

ELIGIBILITY:
All patients undergo upper endoscopy are included after written informed consent is obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient undergoing upper endoscopy after informed consent is obtained
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Kappa coefficient for the intra and inter-rater agreement

CONTACTS AND LOCATIONS:
Overall Officials: Fook Hong Ng, M.D., Principal Investigator — Department of Medicine, Ruttonjee Hospital
Locations (2):
- China (2):
  - Ruttonjee Hospital, Wan Chai, Hong Kong
  - Ruttonjee Hospital, Hong Kong